CLINICAL TRIAL: NCT02853838
Title: Effectiveness of Chest Physiotherapy in Infants Hospitalized With Acute Bronchiolitis SRV (+): a Randomized Controled Trial
Brief Title: Chest Physiotherapy in Infants Between 0 and 12 Months Old With Acute Bronchiolitis SRV(+)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad del Desarrollo (Other)
Collaborators: Hospital Padre Hurtado (Other)
Responsible Party: Principal Investigator, Patricio Gomolan Gonzalez, Lecturer, Universidad del Desarrollo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-84
Record Dates: First submitted 2016-07-22; First posted 2016-08-03 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Bronchiolitis, Viral
Keywords: acute viral bronchiolitis; respiratory syncytial virus; chest physiotherapy
MeSH Terms: conditions — Bronchiolitis, Viral | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolonged slow expiration+provoked coughing+ST (Experimental): Prolonged slow expiration+provoked coughing+Standard Therapy
  Interventions: Other: Prolonged slow expiration+provoked coughing; Other: Standard Therapy
- Manual chest wall vibration+ST (Active Comparator): Manual chest wall vibration+Standard Therapy
  Interventions: Other: Manual chest wall vibration; Other: Standard Therapy

INTERVENTIONS:
Other: Prolonged slow expiration+provoked coughing — Five cycles of prolonged slow expiration and provoked coughing, which will be repeated five times.
  During the prolonged slow expiration, the infant will be in supine while the therapist applies pressure at the same time on the rib cage and abdomen during spontaneous expiration. The pressure is applied slowly during two o three respiratory cycles, only during the final phase of expiration.
  Arms: Prolonged slow expiration+provoked coughing+ST
Other: Manual chest wall vibration — Five cycles of manual chest wall vibrations during 20 seconds each, being repeated five times.
  The manual chest wall vibrations are oscillatory maneuvers applied on the thorax to improve mucociliary clearance of bronchial mucus and ease its removal.
  Arms: Manual chest wall vibration+ST
Other: Standard Therapy — Standard therapy (ST): nasopharyngeal suction, oxygen therapy, fluids administration, 0.5% adrenaline nebulization, and chest physiotherapy.

SUMMARY:
The purpose of this research is to determine the effect of prolonged slow expiration techniques, provoked coughing and standard therapy compared to chest wall manual vibration and standard therapy in infants between 0 and 12 months old with confirmed diagnosis of acute bronchiolitis SRV (+). The effect will be measured on respiratory insufficiency and use of supplementary oxygen.

DETAILED DESCRIPTION:
Bronchiolitis is the main cause of hospital admission for infants under 1 year old in Chile. Currently, approximately 4800 children are admitted to the hospital during the cold season, affecting the health services' effectiveness. The most frequent causal agent is the Respiratory Syncytial Virus (RSV). To date, there is no specific treatment for this disease and only support measures are recommended.

Chest physiotherapy is a support measure that improves the mucociliary clearance and reduces obstruction of the airways.

A clinical trial on the effect of prolonged slow expiration (PSE), chest wall vibrations, and provoked coughing as treatment for bronchiolitis in infants admitted to the hospital found that the subgroup with RSV required oxygen for 10 hours less than the control group. Gomes and Postiaux (2012) reported a 50% decrease on respiratory distress measured by the Wang score when PSE and suction were compared to traditional chest physiotherapy techniques in patients with bronchiolitis RSV(+).

Currently recommendations in Chile suggest chest physiotherapy for outpatients with bronchiolitis, but the guideline does not refer to the case of inpatients. It is proposed to carry out a randomized controlled trial in infants under one year old. The active group will receive standard therapy, PSE, and provoked coughing, while the control group will receive standard therapy and manual chest wall vibrations. The effectiveness of chest physiotherapy will be measured though a clinical score of respiratory distress, hours using supplementary oxygen, vital signs before and after the intervention in both groups during hospital stay. The main outcome is clinical severity score 48 hours after admission.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of bronchiolitis.
* RSV positive in direct immunofluorescence assay.
* Wang clinical severity score ≥ 4 points.

Exclusion Criteria:

* Patients with heart or neurological diseases.
* Previous episodes of wheezing.
* Chronic conditions such as bronchopulmonary dysplasia, immunodeficiency, or congenital diseases.
* Need of mechanical ventilation in Intensive Care Unit
* Contraindication criteria for chest physiotherapy (i.e. Pneumothorax, ribs fractures, hemodynamic instability).
* Patients not receiving supplementary oxygen.

Ages: 15 Days to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 204 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Clinical score of respiratory distress | 48 hours after baseline measurement
  Wang clinical severity score

SECONDARY OUTCOMES:
Hours of supplementary oxygen | 48 hours after baseline measurement
Peripheral blood oxygen level | Baseline, 30 min, 60 min, 120 min,12 hours, 24 hours, 36 hours, and 48 hours.
  Oxygen level or saturation is measured with a pulse oximeter
Heart rate | Baseline, 30 min, 60 min, 120 min,12 hours, 24 hours, 36 hours, and 48 hours.
Respiratory rate | Baseline, 30 min, 60 min, 120 min,12 hours, 24 hours, 36 hours, and 48 hours.
  Wang clinical severity score
wheezing | Baseline, 30 min, 60 min, 120 min,12 hours, 24 hours, 36 hours, and 48 hours.
  Wang clinical severity score
Rib cage retractions | Baseline, 30 min, 60 min, 120 min,12 hours, 24 hours, 36 hours, and 48 hours.
  Wang clinical severity score
General clinical condition | Baseline, 30 min, 60 min, 120 min,12 hours, 24 hours, 36 hours, and 48 hours.
  Wang clinical severity score

OTHER OUTCOMES:
Transfer to high complexity unit | 96 hours
  Categorical variable. Record of number of patients requiring treatment at a higher complexity unit (i.e. ICU)

CONTACTS AND LOCATIONS:
Overall Officials: Patricio Gomolán, Principal Investigator — Universidad del Desarrollo
Locations (1):
- Hospital Padre Hurtado, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available, If journal where report will be published requires to give access to individual patient data

REFERENCES:
- [Derived] Roque-Figuls M, Gine-Garriga M, Granados Rugeles C, Perrotta C, Vilaro J. Chest physiotherapy for acute bronchiolitis in paediatric patients between 0 and 24 months old. Cochrane Database Syst Rev. 2023 Apr 3;4(4):CD004873. doi: 10.1002/14651858.CD004873.pub6. PMID 37010196